CLINICAL TRIAL: NCT02457286
Title: Improving Insulin Resistance to Treat Non-Alcoholic Fatty Liver Disease: A Pilot Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: patients do not want to participate
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, David Bernstein, Chief, Hepatology Center for Liver Diseases, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 13-204
Record Dates: First submitted 2015-05-14; First posted 2015-05-29 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2016-07

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin is being compared to exercise and diet modifications. The study will be incorporating the use of a Fibroscan device (Echosens) at the initial visit and upon completion of the study, which works by measuring shear wave velocity. In this technique, a 50-MHz wave is passed into the liver from a small transducer on the end of an ultrasound probe
  Interventions: Drug: Metformin; Behavioral: Lifestyle modifications; Device: Fibroscan device (Echosens)
- Lifestyle modification (Experimental): The researchers are interested in learning if the addition of metformin to lifestyle modifications is more helpful in treating participants condition or disorder. The study will be incorporating the use of a Fibroscan device (Echosens) at the initial visit and upon completion of the study, which works by measuring shear wave velocity. In this technique, a 50-MHz wave is passed into the liver from a small transducer on the end of an ultrasound probe
  Interventions: Behavioral: Lifestyle modifications; Device: Fibroscan device (Echosens)

INTERVENTIONS:
Drug: Metformin — Although metformin is FDA approved to treat type 2 diabetes, it is not FDA approved for the treatment of NAFLD and is considered investigational for the purpose of this study.
  Other Names: Glucophage
  Arms: Metformin
Behavioral: Lifestyle modifications — Recommendations for lifestyle modification will be based on the Diabetes Prevention Program 2002 (26) and will include recommendations for greater than 150 minutes of physical activity weekly, referrals to group and/or individualized sessions with nutritionists and/or lifestyle coaches as well as educational materials
Device: Fibroscan device (Echosens) — This study will be incorporating the use of a Fibroscan device (Echosens) at the initial visit and upon completion of the study, which works by measuring shear wave velocity.

SUMMARY:
Metformin is being compared to exercise and diet modifications. The researchers are interested in learning if the addition of metformin to lifestyle modifications is more helpful in treating the condition or disorder. Although metformin is FDA approved to treat type 2 diabetes, it is not FDA approved for the treatment of Non-alcoholic fatty liver (NAFLD) and is considered investigational for the purpose of this study.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in the United States and a common cause of unexplained mildly elevated serum aminotransferase levels. NAFLD, initially felt to be benign, is now known to potentially progress to cirrhosis and its complications, including the development of liver cancer. NAFLD is strongly correlated with Type 2 Diabetes, insulin resistance, and the metabolic syndrome (1-6). It is hypothesized that the pathogenesis of hepatic injury in NAFLD is due to insulin resistance and the oxidative stress associated with obesity and metabolic syndrome (7). No adequate medical treatment has been shown to be effective for the treatment of NAFLD. Several studies (8-22) have evaluated the effect of metformin in patients with NAFLD in relation to insulin resistance, Homeostatic Model Assessment Insulin Resistance Index (HOMA-IR) values, aminotransferase levels, liver morphology, and histological improvement with treatment. These studies however have shown discrepant results with relation to aminotransferase levels and only a few studies have been able to evaluate histological improvement with follow-up biopsies. There have been no studies focusing specifically on the pre-diabetic population. These patients who are at an increased risk of progressing to diabetes may exhibit a different response to treatment with metformin than non-diabetic or diabetic patients. All the studies support the fact that metformin has a beneficial effect on improving insulin resistance and decreasing the incidence of metabolic syndrome, but there is no consensus thus far on its influence on NAFLD. The majority of published studies were limited by small sample size. Randomized controlled trials with adequate sample size and of longer duration are needed as well as studies assessing endpoints such as liver morphology and histology. The results of this pilot study are significant in that metformin may be a relatively safe and inexpensive way, in addition to lifestyle modifications, to treat NAFLD. The results of this pilot study will pave the way for the larger power, longer duration study required to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* subjects between ages 18-80
* diagnosed with NAFLD by alanine aminotransferase
* (ALT) levels >1.5x the upper limit of normal with an otherwise nondiagnostic hepatic serology workup, ultrasound evidence, and/or histologically confirmed NAFLD within the past 1 year.
* The upper limit of normal for ALT will be defined as 35 U/L in males and 19 U/L in females

Exclusion Criteria:

* A prior history of diabetes
* Failure to meet criteria for HbA1C screening
* Evidence of hepatic disorders
* Use of insulin or oral hypoglycemic agents
* eGFR <30
* Blood transfusion within past 3 months
* Steroid use in the past 6 months
* Excessive alcohol use (more than 20g per day in women and more than 30g per day in men)
* Acute or unstable congestive heart failure
* Age >80 years old
* Lactic acidosis
* Inability to consent due to cognitive impairment.
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Improvement in NAFLD as measured by ALT levels | 12 Months
  The primary endpoint variable is the improvement in NAFLD after 12 months of treatment, as measured by the change in ALT levels from baseline to the end of a one year follow-up. A decrease of at least 25% from baseline will be considered a clinically relevant response.

SECONDARY OUTCOMES:
Incidence of metabolic syndrome (insulin resistance) | 12 months
  The study will be using measurements of BMI, waist circumference, blood pressure, lipids and fasting blood glucose levels to assess insulin resistance.
Incidence of NAFLD fibrosis scores after 12 months of treatment as measured by Fibroscan | 12 months
  A NAFLD Fibrosis Score (28), a noninvasive scoring system for liver fibrosis in patients with NAFLD, can be calculated and potentially used to assess for histologic improvement with metformin, which thus far has never been assessed.

CONTACTS AND LOCATIONS:
Overall Officials: David Bernstein, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore Hospital, Manhasset, New York, United States

REFERENCES:
- [Result] Ortiz-Lopez C, Lomonaco R, Orsak B, Finch J, Chang Z, Kochunov VG, Hardies J, Cusi K. Prevalence of prediabetes and diabetes and metabolic profile of patients with nonalcoholic fatty liver disease (NAFLD). Diabetes Care. 2012 Apr;35(4):873-8. doi: 10.2337/dc11-1849. Epub 2012 Feb 28. PMID 22374640
- [Result] Arase Y, Suzuki F, Ikeda K, Kumada H, Tsuji H, Kobayashi T. Multivariate analysis of risk factors for the development of type 2 diabetes in nonalcoholic fatty liver disease. J Gastroenterol. 2009;44(10):1064-70. doi: 10.1007/s00535-009-0091-1. Epub 2009 Jun 17. PMID 19533014
- [Result] Bedogni G, Miglioli L, Masutti F, Tiribelli C, Marchesini G, Bellentani S. Prevalence of and risk factors for nonalcoholic fatty liver disease: the Dionysos nutrition and liver study. Hepatology. 2005 Jul;42(1):44-52. doi: 10.1002/hep.20734. PMID 15895401
- [Result] Adams LA, Waters OR, Knuiman MW, Elliott RR, Olynyk JK. NAFLD as a risk factor for the development of diabetes and the metabolic syndrome: an eleven-year follow-up study. Am J Gastroenterol. 2009 Apr;104(4):861-7. doi: 10.1038/ajg.2009.67. Epub 2009 Mar 17. PMID 19293782
- [Result] Nar A, Gedik O. The effect of metformin on leptin in obese patients with type 2 diabetes mellitus and nonalcoholic fatty liver disease. Acta Diabetol. 2009 Jun;46(2):113-8. doi: 10.1007/s00592-008-0067-2. Epub 2008 Oct 7. PMID 18839053
- [Result] Lidofsky SD. Nonalcoholic fatty liver disease: diagnosis and relation to metabolic syndrome and approach to treatment. Curr Diab Rep. 2008 Feb;8(1):25-30. doi: 10.1007/s11892-008-0006-1. PMID 18366995